CLINICAL TRIAL: NCT00513084
Title: Moderators and Mediators of Physical Activity, Body Weight, and Body Composition Change During Obesity Treatment in Women
Brief Title: Promotion of Exercise and Health in Obesity
Acronym: PESO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Lisbon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCT-POCI/DES/57705/2004
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-07

CONDITIONS: Obesity
Keywords: Behavioral,; Self-Determination Theory,; Motivational Interviewing,; Exercise, Physical Activity,; Motivation,; Moderators,; Mediators,; Predictors,; Weight
MeSH Terms: conditions — Obesity; Behavior; Motor Activity; Body Weight | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SDT Intervention (Experimental): This arm will follow main experimental intervention, as described elsewhere
  Interventions: Behavioral: SDT and Motivational Interviewing in Obesity Treatment
- Comparison Group (No Intervention): Comparison Group receiving standard care health promotion intervention

INTERVENTIONS:
Behavioral: SDT and Motivational Interviewing in Obesity Treatment — Thirty group sessions, designed to follow SDT, covering PA, eating/nutrition, body image, and other cognitive-behavioral contents. Central to the intervention are improving autonomy, intrinsic motivation, and self-regulation of behavior change. Accepting ambivalence for change, rolling with resistance, and developing discrepancy were used throughout the program, with an emphasis on promoting intrinsic, self-regulated motivation for exercise and weight control.
  Other Names: GI: Intervention Group
  Arms: SDT Intervention

SUMMARY:
The primary objectives of this randomized clinical trial are a) to implement and test the impact of a 1-year lifestyle obesity treatment program based on Self-Determination Theory on 3-year change in physical activity and motivation for exercise/physical activity, body weight and fat, and selected eating variables, b) to identify behavioral and psychosocial theory-based moderators or mediators of primary outcomes, especially physical activity and body weight.

DETAILED DESCRIPTION:
Obesity and sedentary lifestyles are worldwide threats to public health but feasible and effective strategies to tackle these problems are scarce. The identification of variables that explain why only a sub-group of overweight persons succeeds at increasing physical activity and achieving long-term weight control is a key research topic in exercise and sports sciences. Subjects are 260 healthy women (BMI, 25 to 40 kg/m2), aged between 25 and 50 years, premenopausal, of whom half receive the treatment intervention, the remaining being randomly assigned to a control group at baseline. This RCT consists of a 1-year intervention plus a 2-year no contact follow-up period. The intervention group attended 30 weekly group sessions, designed to follow SDT basic tenets, covering PA, eating/nutrition, body image, and other cognitive and behavioral contents. Central to the intervention model are autonomy, intrinsic motivation, and self-regulation of behavior change. Autonomy-supportive treatment climate and internal causality orientations are predicted to enhance autonomous regulation, perceived competence, and intrinsic motivation for the targeted behaviors, resulting in lasting behavioral and body weight changes. The intervention was designed to follow SDT, with an emphasis on promoting intrinsic, self-regulated motivation for exercise and weight control. The control group received a general health education curriculum based on several 3- to 6-week long educational topics (e.g. food safety, stress management, self-care, body image, and others). Results are expected to contribute to a better understanding of how individual characteristics, particularly those related to physical activity and exercise influence success, better screening/readiness testing procedures, improved matching of interventions to participants, and lower rates of attrition and unsuccessful weight loss attempts.

ELIGIBILITY:
Inclusion Criteria:

* female (25-50 years old)
* pre-menopausal
* BMI between 25 and 40 kg/m2
* willing to attend weekly meetings (during 1 year)
* willing to not participate in other formal or informal weight loss program during the first year of the study (intervention group only).

Exclusion Criteria:

* major/chronic illness
* taking (or having taken in the previous year) medication known to interfere with body weight regulation, including anti-depressive medication

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 259 (Actual)
Dates: Start 2004-07; Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Primary outcomes are physical activity/exercise and body weight/ composition. Physical activity is assessed by accelerometry and standardized interview/questionnaire methods. Body composition is assessed by DXA | baseline, 4, 12, 16, 24 and 36 months

SECONDARY OUTCOMES:
Dietary Intake, psychosocial SDT-based mediators | baseline, 4, 12,16, 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J Teixeira, PhD, Principal Investigator — Faculty of Human Movement, Technical University of Lisbon; Luis B Sardinha, PhD, Principal Investigator — Faculty of Human Movement, Technical University of Lisbon
Locations (1):
- Faculty of Human Movement, Technical University of Lisbon, Lisbon, Estrada Da Costa, Portugal

REFERENCES:
- [Result] Minderico CS, Silva AM, Fields DA, Branco TL, Martins SS, Teixeira PJ, Sardinha LB. Changes in thoracic gas volume with air-displacement plethysmography after a weight loss program in overweight and obese women. Eur J Clin Nutr. 2008 Mar;62(3):444-50. doi: 10.1038/sj.ejcn.1602709. Epub 2007 Mar 28. PMID 17392701
- [Result] Teixeira PJ, Going SB, Houtkooper LB, Cussler EC, Metcalfe LL, Blew RM, Sardinha LB, Lohman TG. Exercise motivation, eating, and body image variables as predictors of weight control. Med Sci Sports Exerc. 2006 Jan;38(1):179-88. doi: 10.1249/01.mss.0000180906.10445.8d. PMID 16394972
- [Derived] Jorge R, Santos I, Tomas R, Silva MN, Carraca EV, Teixeira VH, Teixeira PJ. Behavioural and psychological pretreatment predictors of short- and long-term weight loss among women with overweight and obesity. Eat Weight Disord. 2020 Oct;25(5):1377-1385. doi: 10.1007/s40519-019-00775-9. Epub 2019 Sep 13. PMID 31520301
- [Derived] Carraca EV, Markland D, Silva MN, Coutinho SR, Vieira PN, Minderico CS, Sardinha LB, Teixeira PJ. Physical activity predicts changes in body image during obesity treatment in women. Med Sci Sports Exerc. 2012 Aug;44(8):1604-12. doi: 10.1249/MSS.0b013e31824d922a. PMID 22330022
- [Derived] Silva MN, Markland D, Carraca EV, Vieira PN, Coutinho SR, Minderico CS, Matos MG, Sardinha LB, Teixeira PJ. Exercise autonomous motivation predicts 3-yr weight loss in women. Med Sci Sports Exerc. 2011 Apr;43(4):728-37. doi: 10.1249/MSS.0b013e3181f3818f. PMID 20689448
- [Derived] Teixeira PJ, Silva MN, Coutinho SR, Palmeira AL, Mata J, Vieira PN, Carraca EV, Santos TC, Sardinha LB. Mediators of weight loss and weight loss maintenance in middle-aged women. Obesity (Silver Spring). 2010 Apr;18(4):725-35. doi: 10.1038/oby.2009.281. Epub 2009 Aug 20. PMID 19696752
- [Derived] Silva MN, Markland D, Minderico CS, Vieira PN, Castro MM, Coutinho SR, Santos TC, Matos MG, Sardinha LB, Teixeira PJ. A randomized controlled trial to evaluate self-determination theory for exercise adherence and weight control: rationale and intervention description. BMC Public Health. 2008 Jul 9;8:234. doi: 10.1186/1471-2458-8-234. PMID 18613959